CLINICAL TRIAL: NCT02200250
Title: Long Term Outcomes of Patients Undergoing Endoscopic Resection of Barrett's Oesophagus (BO) With High Grade Dysplasia (HGD) and Early Adenocarcinoma
Brief Title: Long Term Barrett's Endoscopic Mucosal Resection Study
Acronym: CBE
Status: Withdrawn | Type: Observational
Why Stopped: Study abandoned
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2013/10/6.2(3838)QA
Record Dates: First submitted 2014-07-17; First posted 2014-07-25 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Barretts Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Post Barretts Excision: Patients who have undergone an EMR for Barretts Oesophagus

SUMMARY:
Analysis of long term outcomes of patients undergoing endoscopic mucosal resection for Barrett's oesophagus with high grade dysplasia and/or early intramucosal carcinoma (IMC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* Have or have had Barrett's Oesophagus

Exclusion Criteria:

* Do not have Barrett's Oesophagus
* Have not had Barrett's Oesophagus resected at Westmead Hospital

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have or have had Barrett's Oesophagus with high grade dysplasia or adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Reviewing patients symptoms following resection | up to 3 years
  Patients will be contacted via phone and will be required to answer questions over the phone. Health questionnaires may also be sent at the patients request to complete and post back.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia